CLINICAL TRIAL: NCT02817074
Title: MIND Diet Intervention to Prevent Alzheimer's Disease
Brief Title: MIND Diet Intervention and Cognitive Decline
Acronym: MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Brigham and Women's Hospital (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lisa L. Barnes, PhD, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AG051641 (NIH); 1R01AG052583-01 (NIH)
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Cognitive Decline; Dementia; Alzheimer Disease; Vascular Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIND Diet +Weight loss (Active Comparator): 3-year intervention of dietary counseling to adhere to the MIND diet plus reduce calorie intake by 250 kcal /day for mild weight loss
  Interventions: Behavioral: MIND Diet; Behavioral: Mild Weight Loss
- Usual Diet + Weight Loss (Placebo Comparator): 3-year intervention of usual diet + counseling to reduce calorie intake by 250 kcal/day for mild weight loss
  Interventions: Behavioral: Mild Weight Loss

INTERVENTIONS:
Behavioral: MIND Diet — 3-year dietary counseling to adhere to the MIND diet and for mild weight loss
  Arms: MIND Diet +Weight loss
Behavioral: Mild Weight Loss — 3-year dietary counseling to reduce calorie intake by 250 kcal/day for mild weight loss

SUMMARY:
Phase III randomized controlled trial designed to test the effects of a 3-year intervention of the MIND diet (Mediterranean-DASH Intervention for Neurodegenerative Delay) on cognitive decline and brain neurodegeneration among 600 individuals 65+ years without cognitive impairment who are overweight and have suboptimal diets.

DETAILED DESCRIPTION:
Mediterranean-DASH Diet Intervention for Neurodegenerative Delay (MIND) is a Phase III randomized controlled trial designed to test the effects of a 3-year intervention of a hybrid of the Mediterranean and DASH diets, called MIND, on cognitive decline among 600 individuals 65+ years without cognitive impairment who are overweight and have suboptimal diets. The proposed MIND diet is a hybrid of the Mediterranean and DASH diets but with selected modifications based on the most compelling evidence in the diet-dementia field. The MIND diet has the same basic components of the DASH and Mediterranean diets, such as emphasis on natural plant-based foods and limited animal and high saturated fat foods, but uniquely specifies green leafy vegetables and berries as well as food component servings that reflect the nutrition-dementia evidence. The trial will employ a parallel group design comparing the effects on cognitive outcomes of the MIND intervention diet plus mild caloric restriction for weight loss to the control diet, usual diet with mild caloric restriction for weight loss. Biological effects of the MIND diet will be assessed by measurement of brain macro- and micro-structural integrity in 300 randomly selected participants. Other biochemical markers will be assessed in the entire cohort of 600 participants, including: plasma Abeta 42/Abeta 40, brain-derived neurotrophic factor (BDNF) and plasma markers of oxidative stress and inflammation. In addition, the trial will examine potential effect mediators and modifiers by a number of cardiovascular risk factors, AD biomarkers, and biological mechanisms. The proposed study has two clinical sites, one in Chicago (Rush University) and one in Boston (Harvard University), and centralized laboratories for data coordinating and analyses (Brigham & Women's Hospital), neuroimaging analyses (Rush University), and specialized laboratories for tissue biochemical analyses.

ELIGIBILITY:
Inclusion Criteria:

* family history of dementia
* BMI >=25
* suboptimal diet

Exclusion Criteria:

* heavy alcohol use
* severe illness
* cognitively impaired
* psychiatric illness

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 604 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in global cognitive function (composite score) | 3 years
  Global cognitive function assessment is based on a battery of 12 cognitive tests [1. Word list Memory; 2. Word List Recall; 3. Word List Recognition; 4. Logical Memory (East Boston Story Immediate Recall); 5. Logical Memory (East Boston Story Delayed Recall); 6. Verbal Fluency; 7. Multilingual Naming Test; 8. Trail A; 9. Trail B; 10. Flanker Inhibitory Control; 11. Oral Symbol Digit Modalities Test; and 12. Pattern Comparison. Individual test scores will be summarized by calculating the z-score for each test based on the mean and standard deviation of the sample distribution - averaging z-scores across tests will yield a composite score for global cognitive function. Cognitive function will be assessed at the baseline, 6, 12, 24, and 36 months to determine the time-course of cognitive change.
Change in specific cognitive domains | 3 years
  Change in specific cognitive domains: episodic memory, semantic memory, perceptual speed, and executive function

SECONDARY OUTCOMES:
Change in brain MRI total brain /intracranial volume (cubic centimeters) and hippocampal/intracranial volume (cubic centimeters) | 3 years
  Changes in brain MRI-derived normalized measures of total brain volume (cubic centimeters) and hippocampal volume (cubic centimeters) and white/gray matter, segmented gray matter regions, white matter lesions, and thickness of segmented cortical regions.

OTHER OUTCOMES:
Exploratory aim 1: Incidence of cardiovascular disease | 3 years
  To evaluate the role of MIND diet on the risk of incident cardiovascular disease. Cardiovascular disease is defined as the presence of coronary heart disease, cerebrovascular disease, and/or heart failure.
Exploratory aim 2a: Blood pressure | 3 years
  To evaluate the role of MIND diet on the change of systolic and diastolic blood pressure (mmHg) from the baseline to 6, 12, 24, and 36 months
Exploratory aim 2b: Total cholesterol | 3 years
  To evaluate the role of MIND diet on the change of total cholesterol (mg/dL), in plasma from the baseline to 3 and 36 months.
Exploratory aim 2c: Low-density lipoprotein (LDL) | 3 years
  To evaluate the role of MIND diet on the change of LDL (mg/dL) in plasma from the baseline to 3 and 36 months.
Exploratory aim 2d: High-density lipoprotein (HDL) | 3 years
  To evaluate the role of MIND diet on the change of HDL (mg/dL) in plasma from the baseline to 3 and 36 months.
Exploratory aim 2e: Hemoglobin A1c (HbA1c) | 3 years
  To evaluate the role of MIND diet on the change of HbA1c levels in plasma from the baseline to 3 and 36 months.
Exploratory aim 3: Plasma amyloid beta (Abeta) | 3 years
  To evaluate the role of MIND diet on the change of plasma Abeta 40 (pg/ml), Abeta42 (pg/ml), and ratio Abeta40/Abeta42 from the baseline to 3 and 36 months.
Exploratory aim 4a: C-Reactive Protein (CRP) | 3 years
  To evaluate the role of MIND diet on the change of CRP (mg/L) levels in plasma from the baseline to 3 and 36 months.
Exploratory aim 4b: Interleukin 6 (IL-6) | 3 years
  To evaluate the role of MIND diet on the change of plasma IL-6 (pg/mL) from the baseline to 3 and 36 months.
Exploratory aim 4c: Oxidized LDL | 3 years
  To evaluate the role of MIND diet on the change of oxidized LDL (mg/dl) in plasma from the baseline to 3 and 36 months.
Exploratory aim 4d: Estimated glomerular filtration rate (eGFR) | 3 years
  To evaluate the role of MIND diet on the change of eGFR (mg/dL) from the baseline to 3 and 36 months.
Exploratory aim 4e: Brain-derived neurotrophic factor | 3 years
  To evaluate the role of MIND diet on the change of plasma Brain-derived neurotrophic factor (pg/mL) from the baseline to 3 and 36 months.
Exploratory aim 4f: Adiponectin | 3 years
  To evaluate the role of MIND diet on the change of plasma adiponectin (mg/L) levels from the baseline to 3 and 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Barnes, Ph.D., Principal Investigator — Rush University
Locations (2):
- United States (2):
  - Rush University, Chicago, Illinois
  - Harvard School of Public Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Electronic data will be made available after trial completion

REFERENCES:
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimers Dement. 2015 Sep;11(9):1007-14. doi: 10.1016/j.jalz.2014.11.009. Epub 2015 Feb 11. PMID 25681666
- [Derived] Halloway S, Aggarwal NT, Arfanakis K, Sacks FM, Barnes LL, Dhana K. Effect modifiers of the MIND diet for cognition in older adults: The MIND diet trial. Alzheimers Dement. 2025 Oct;21(10):e70731. doi: 10.1002/alz.70731. PMID 41058007
- [Derived] Dhana K, Aggarwal NT, Voigt RM, Ventrelle J, Rajan KB, Kaddurah-Daouk R, Marcovina SM, Liu X, Agarwal P, Tangney C, Arfanakis K, Sacks FM, Barnes LL. Effect of weight loss through dietary interventions on cardiometabolic health in older adults. Int J Obes (Lond). 2025 Dec;49(12):2503-2510. doi: 10.1038/s41366-025-01902-6. Epub 2025 Oct 3. PMID 41044190
- [Derived] Liu X, Sacks FM, Beck T, Tangney CC, Willett WC, Yassine H, Dhana K, Aggarwal NT, Rajan KB, Barnes LL. Apolipoprotein E epsilon4-dependent associations between carotenoids and cognitive decline: Findings from the MIND (Mediterranean-DASH Intervention for Neurodegenerative delay) randomized controlled trial. Am J Clin Nutr. 2025 Nov;122(5):1289-1297. doi: 10.1016/j.ajcnut.2025.08.012. Epub 2025 Aug 27. PMID 40876538
- [Derived] Barnes LL, Dhana K, Liu X, Carey VJ, Ventrelle J, Johnson K, Hollings CS, Bishop L, Laranjo N, Stubbs BJ, Reilly X, Agarwal P, Zhang S, Grodstein F, Tangney CC, Holland TM, Aggarwal NT, Arfanakis K, Morris MC, Sacks FM. Trial of the MIND Diet for Prevention of Cognitive Decline in Older Persons. N Engl J Med. 2023 Aug 17;389(7):602-611. doi: 10.1056/NEJMoa2302368. Epub 2023 Jul 18. PMID 37466280
- [Derived] Liu X, Dhana K, Furtado JD, Agarwal P, Aggarwal NT, Tangney C, Laranjo N, Carey V, Barnes LL, Sacks FM. Higher circulating alpha-carotene was associated with better cognitive function: an evaluation among the MIND trial participants. J Nutr Sci. 2021 Aug 16;10:e64. doi: 10.1017/jns.2021.56. eCollection 2021. PMID 34527222
- [Derived] Lefevre-Arbogast S, Dhana K, Aggarwal NT, Zhang S, Agarwal P, Liu X, Laranjo N, Carey V, Sacks F, Barnes LL, Arfanakis K. Vitamin D Intake and Brain Cortical Thickness in Community-Dwelling Overweight Older Adults: A Cross-Sectional Study. J Nutr. 2021 Sep 4;151(9):2760-2767. doi: 10.1093/jn/nxab168. PMID 34113981
- [Derived] Halloway S, Dhana K, Desai P, Agarwal P, Holland T, Aggarwal NT, Evers J, Sacks FM, Carey VJ, Barnes LL. Free-Living Standing Activity as Assessed by Seismic Accelerometers and Cognitive Function in Community-Dwelling Older Adults: The MIND Trial. J Gerontol A Biol Sci Med Sci. 2021 Oct 13;76(11):1981-1987. doi: 10.1093/gerona/glab106. PMID 33835152
- [Derived] Liu X, Morris MC, Dhana K, Ventrelle J, Johnson K, Bishop L, Hollings CS, Boulin A, Laranjo N, Stubbs BJ, Reilly X, Carey VJ, Wang Y, Furtado JD, Marcovina SM, Tangney C, Aggarwal NT, Arfanakis K, Sacks FM, Barnes LL. Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) study: Rationale, design and baseline characteristics of a randomized control trial of the MIND diet on cognitive decline. Contemp Clin Trials. 2021 Mar;102:106270. doi: 10.1016/j.cct.2021.106270. Epub 2021 Jan 9. PMID 33434704